CLINICAL TRIAL: NCT00627978
Title: Phase II Study of Ixabepilone in Patients With Metastatic Breast Cancer and a Prospective Evaluation of Its Effects on the Ultrastructure of Neurons
Brief Title: Phase II Study of Ixabepilone in Metastatic Breast Cancer and Its Effects on the Ultrastructure of Neurons
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0707009284
Record Dates: First submitted 2008-02-22; First posted 2008-03-04 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Breast Cancer
Keywords: breast
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ixabepilone (Experimental): Participants are treated with Ixabepilone.
  Interventions: Drug: ixabepilone
- Control (No Intervention)

INTERVENTIONS:
Drug: ixabepilone — ixabepilone 40 mg/m2 Q3w over 3 hours
  Arms: Ixabepilone

SUMMARY:
Primary Objectives

* Assess ultrastructure changes in dermal myelinated nerves of patients who receive ixabepilone chemotherapy
* Detailed characterization of peripheral neuropathy in patients who receive ixabepilone

Secondary Objectives

* Clinical benefit rate
* Time to progression ( TTP)
* Toxicity
* Exploratory studies:

  * Relation of MDR 1 and TRKA polymorphisms to evolution of ultrastructural neurologic changes observed in neurons.
  * Relation of NGF, IL8, and IL10 to the development of clinical symptoms and ultrastructural changes in neurons.

DETAILED DESCRIPTION:
Eligible patient population:

* Stage 4 breast cancer
* Resolution from toxicity of prior therapy to ≤ CTC grade 1 ( except alopecia)
* No limit on prior number of therapies to treat cancer
* Adequate organ function
* Life expectancy greater than 3 months

Treatment: ixabepilone 40 mg/m2 Q3w over 3 hours

Evaluation on Study:

I. Efficacy evaluation:

* Baseline CT chest, abdomen and pelvis and bone scan within 4 weeks of starting therapy
* Evaluation of disease every 2 cycles of chemotherapy
* Ongoing toxicity evaluation using NCI CTC 3.

II. Neurological evaluation:

* Detailed neurologic exam using Neuropathy Assessment Instrument (represents a standard neurological exam)
* Serum NGF, IL 8,10, prior to starting therapy and prior to each cycle of ixabepilone
* DNA for assessment of TRK A and MDR1 polymorphisms
* Punch biopsy of skin prior to starting therapy and after every 2 cycles. Laboratory evaluation of peripheral nerve biopsies will be conducted at Rockefeller University under the direction of Dr. Carlson in Dr. Strickland's Lab.

ELIGIBILITY:
Inclusion Criteria

* Ability to understand and the willingness to sign a written informed consent document.
* Histologic or cytologic diagnosis of adenocarcinoma originating in the breast.
* Evidence that the cancer is metastatic or locally advanced and not curable by local measures (i.e., surgery, radiation).

NOTE: There is no limit on number of prior chemotherapy regimens received.

* Karnofsky performance status (KPS) score of 70 - 100; (Appendix 1).
* Life expectancy of at least 12 weeks.
* Adequate recovery of drug related toxicities from prior systemic therapy (recovery to < = Grade 1 except for Grade 2 fatigue and alopecia).
* Adequate recovery from recent surgery and radiation therapy. At least one week must have elapsed from the time of a minor surgery and/or focal/palliative radiation therapy; at least 3 weeks for major surgery and other radiation therapy.
* Women or Men, age > = 18 years.
* Patients must have normal organ and marrow function as defined below:

  * Hematologic function with absolute neutrophils ≥ 1,500/mm3 and/or platelets > 125,000/mm3
  * Hepatic function with serum bilirubin less than 1.5 times the upper institutional limits of normal, ALT ≤ 2.5 times the upper institutional limits of normal (≤ 5 times the upper institutional limits of normal if documented hepatic metastases are present)
  * Renal function with serum creatinine ≤ 1.5 times the upper limit of normal
* Women of childbearing potential (WOCBP) and men with partners who are of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study in such a manner that the risk of pregnancy is minimized.

WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea > = 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL). Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential.

- WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication.

Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria

* Patients with known and active brain and/or leptomeningeal metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* CTC Grade 2 or greater neuropathy (motor or sensory) at study entry.
* Prior treatment with ixabepilone.
* Serious intercurrent infections, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy, including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known history of HIV infection.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other concurrent chemotherapy, hormonal therapy, immunotherapy regimens or radiation therapy, standard or investigational.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ixabepilone.
* Known prior severe hypersensitivity reactions to agents containing CremophorEL.
* Patients may not be receiving any prohibited therapies and/or medications.
* Pregnant and lactating women are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Vahdat, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: No treatment with Ixabepilone
Period: Overall Study
Arm/Group | Ixabepilone | Control
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Participants receive no intervention.
- Total: Total of all reporting groups
Arm/Group | Ixabepilone | Control | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years] | 55.8 [39 to 70] | 51 [35 to 63] | 54.4 [35 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Axons With Abnormal Morphology
Description: Digital photographs for morphometry were captured at a magnification of 8000-16,000x and the photos were uploaded onto an imaging platform of transmission electron microscope (iTEM) (Olympus, Mu¨nster, Germany). The figures were enlarged by 50%, and an individual linear array was used to measure the axonal diameter (cross-sectional area) and the number of unmyelinated axons per Remak Schwann cell was enumerated according to the established methodology.
Time Frame: Baseline and Over 7 cycles of treatment, approximately 21 weeks
Measure: Number; unit: percentage of axons
Arm/Group | Ixabepilone | Control
Number analyzed (Participants) | 10 | 5
percentage of axons
  Axons grade 0 (normal) or 1 morphology baseline | 52 | 82
  Axons grade 0 (normal) or 1 morphology Cycle 7 | 2 | NA — Treatment was not given to the control arm so no value is available for post-7 cycles of treatment
  Axons grade 3 or 4 morphology baseline | 24 | 15.5
  Axons grade 3 or 4 morphology Cycle 7 | 79 | NA — Treatment was not given to the control arm so no value is available for post-7 cycles of treatment

ADVERSE EVENTS:
Description: Serious and Other [Not Including Serious] Adverse Events were not collected/assessed.
Groups:
- Control: Participants are not treated with Ixabepilone.
Arm/Group | Ixabepilone | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No